CLINICAL TRIAL: NCT01180699
Title: A Randomized Controlled Trial Comparing Intradermal vs. Intramuscular Trivalent Inactivated Influenza Vaccine in Adult Solid Organ Transplant Recipients
Brief Title: Intradermal Versus Intramuscular Trivalent Influenza Vaccine in Adult Solid Organ Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Deepali Kumar, Assistant Professor of Medicine, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KUOA-02
Record Dates: First submitted 2010-06-10; First posted 2010-08-12 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Influenza Vaccine
Keywords: adult solid organ transplant patients
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- influenza vaccine - intradermal (Experimental): intradermal versus intramuscular
  Interventions: Biological: Influenza vaccine: Vaxigrip or Fluviral and Intanza
- influenza vaccine - intramuscular (Active Comparator)
  Interventions: Biological: Influenza vaccine: Vaxigrip or Fluviral and Intanza

INTERVENTIONS:
Biological: Influenza vaccine: Vaxigrip or Fluviral and Intanza — Patients will be randomized to receive either one intradermal dose of 0.1 mL or one intramuscular injection of 0.5 mL of the standard influenza vaccine in the deltoid muscle of the nondominant arm.

SUMMARY:
Influenza virus is an important cause of morbidity in the transplant population and can lead to viral and bacterial pneumonia and contribute to the development of rejection. Although the annual influenza vaccine is recommended for transplant patients, studies have shown that a single intramuscular dose has poor immunogenicity. There are no studies that define the effect of intradermal doses in this population. We plan to study the immunogenicity of two different administration routes of the influenza vaccine in 200 solid organ transplant patients during the 2010-2011 season. Patients will be randomized to receive influenza vaccine either intradermally or intramuscularly. We hypothesize that the patients who receive the intradermal influenza vaccine will significantly reach a higher response to the vaccine. This study advances research on the prevention of serious viral infections in transplant recipients. Results from this study have the potential to directly improve patient care. If the use of the intradermal influenza vaccine is successful, this strategy may lead to a significant reduction in burden of disease, hospitalizations, and long-term morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 59,
* Greater than 3 months post-transplant,
* Any solid organ transplant (kidney, liver, heart, lung, pancreas, intestinal or combinations of the aforementioned organs)

Exclusion Criteria:

* Has already received influenza vaccination for 2010-2011 season;
* Egg allergy,
* Previous life-threatening reaction to influenza vaccine (i.e. Guillain Barre Syndrome),
* Ongoing therapy for rejection,
* Febrile illness in the past two weeks,
* Unable to provide informed consent,
* Unable to comply with study protocol

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 229 (Actual)
Dates: Start 2010-10; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate: serological response with a four-fold or greater increase in HI antibody titers to an antigen | 4 weeks

SECONDARY OUTCOMES:
Local and systemic adverse events to vaccination | 24 hours, 48 hours and 7 days after each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Kumar, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada